CLINICAL TRIAL: NCT00591253
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of TAK-491 in Black Subjects With Essential Hypertension
Brief Title: Efficacy and Safety of Azilsartan Medoxomil in African American Participants With Essential Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sr. VP, Clinical Science, Takeda Global Research & Development Center, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-491-011; U1111-1113-8925 (Registry Identifier: WHO)
Record Dates: First submitted 2007-12-27; First posted 2008-01-11 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Hypertension
Keywords: Blood pressure; blood pressure monitoring ambulatory; Drug Therapy
MeSH Terms: conditions — Hypertension | interventions — azilsartan medoxomil; azilsartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Azilsartan Medoxomil 40 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Azilsartan Medoxomil 80 mg QD (Experimental)
  Interventions: Drug: Azilsartan medoxomil
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azilsartan medoxomil — Azilsartan medoxomil 40 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 40 mg QD
Drug: Azilsartan medoxomil — Azilsartan medoxomil 80 mg, tablets, orally, once daily for up to 6 weeks.
  Other Names: TAK-491; Edarbi
  Arms: Azilsartan Medoxomil 80 mg QD
Drug: Placebo — Azilsartan medoxomil placebo-matching tablets, orally, once daily for up to 6 weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of azilsartan medoxomil compared to placebo, once daily (QD), in African-American participants with essential hypertension.

DETAILED DESCRIPTION:
Hypertension affects approximately 50 million individuals in the United States. As the population ages, the prevalence of hypertension will continue to increase if broad and effective preventive measures are not implemented. According to the World Health Organization, hypertension is the most common attributable cause of preventable death in developed nations, as uncontrolled hypertension greatly increases the risk of cardiovascular disease, cerebrovascular disease, and renal failure. Despite the availability of antihypertensive treatments, hypertension remains inadequately controlled; only about one third of patients continue to maintain control successfully.

A major component of blood pressure regulation is the renin-angiotensin-aldosterone system, a system of hormone-mediated feedback interactions that results in the relaxation or constriction of blood vessels in response to various stimuli. Angiotensin II, a polypeptide hormone, is formed from angiotensin I in a reaction catalyzed by angiotensin-converting enzyme as part of the renin-angiotensin-aldosterone system. Angiotensin II is the principal pressor agent of the renin-angiotensin-aldosterone system with a myriad of effects on the cardiovascular system and on electrolyte homeostasis.

In the United States, a disproportionate number of African-Americans have hypertension compared to age-matched non-Hispanic Caucasians and Mexican Americans. Earlier onset and greater severity of hypertension in African-Americans contribute to greater target organ damage and may be a factor in shorter life expectancy in this population compared to Caucasian-Americans. Although genetic factors have been invoked to explain these racial differences, environmental factors probably play a more important role. Improved management of hypertension through both lifestyle intervention and pharmacotherapy, including combination therapy, are necessary to achieve target blood pressure in African Americans.

Takeda Global Research & Development Center, Inc. is developing TAK-491 (azilsartan medoxomil) to treat patients with essential hypertension. Azilsartan medoxomil is a prodrug that is hydrolyzed to the active moiety, TAK-536 (azilsartan), which is a selective antagonist of the angiotensin II type 1 receptor subtype.

This study is being conducted to evaluate the effectiveness and safety of oral azilsartan medoxomil compared with placebo in African-American participants with essential hypertension. Participation in this study is anticipated to be approximately 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The participant has essential hypertension (defined as sitting trough clinic systolic blood pressure between 150 and 180 mm Hg, inclusive at Day -1) and 24-hour mean systolic blood pressure 130-170 mm Hg, inclusive, at Day 1.
2. Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
3. Clinical laboratory evaluations within the reference range for the testing laboratory unless the results are deemed not clinically significant for inclusion into this study by the investigator.
4. Willing to discontinue current antihypertensive medication.

Exclusion Criteria:

1. Has sitting trough clinic diastolic blood pressure greater than 114 mm Hg.
2. Baseline 24 hour ambulatory blood pressure monitor reading of insufficient quality.
3. Hypersensitive to angiotensin II receptor blockers.
4. History of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebrovascular accident, or transient ischemic attack.
5. Clinically significant cardiac conduction defects.
6. Hemodynamically significant left ventricular outflow obstruction due to aortic valvular disease.
7. Secondary hypertension of any etiology.
8. Non-compliant with study medication during run-in period.
9. Severe renal dysfunction or disease (based on calculated creatinine clearance less than 30 mL/min/1.73 m2) at Screening.
10. Known or suspected unilateral or bilateral renal artery stenosis.
11. History of drug abuse or a history of alcohol abuse within the past 2 years.
12. Previous history of cancer that has not been in remission for at least 5 years prior to the first dose of study drug.
13. Type 1 or poorly controlled type 2 diabetes mellitus.
14. Alanine aminotransferase level of greater than 2.5 times the upper limit of normal, active liver disease, or jaundice.
15. Hyperkalemia.
16. Upper arm circumference less than 24 cm or greater than 42 cm.
17. Works night (3rd) shift.
18. Currently is participating in another investigational study or has participated in an investigational study within 30 days prior to randomization.
19. Any other serious disease or condition at Screening (or Randomization) that would compromise participant safety, might affect life expectancy, or make it difficult to successfully manage and follow the participant according to the protocol.
20. Randomized in a previous azilsartan medoxomil study.
21. Is required to take or continues taking any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Executive Medical Director Clinical Science, Study Director — Takeda
Locations (64):
- United States (60):
  - Alabaster, Alabama
  - Huntsville, Alabama
  - Tempe, Arizona
  - Freemont, California
  - Garden Grove, California
  - Long Beach, California
  - Riverside, California
  - Sacramento, California
  - San Diego, California
  - Whittier, California
  - Newark, Delaware
  - Hialeah, Florida
  - Hollywood, Florida
  - Miami, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Waycross, Georgia
  - Chicago, Illinois
  - Avon, Indiana
  - Elkhart, Indiana
  - Indianapolis, Indiana
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Ann Arbor, Michigan
  - Bingham Farms, Michigan
  - Southfield, Michigan
  - Florissant, Missouri
  - Brooklyn, New York
  - Hickory, North Carolina
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Shelby, North Carolina
  - Akron, Ohio
  - Centerville, Ohio
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Willoughby Hills, Ohio
  - Zanesville, Ohio
  - Oklahoma City, Oklahoma
  - Downingtown, Pennsylvania
  - Jenkintown, Pennsylvania
  - Anderson, South Carolina
  - Charleston, South Carolina
  - Simpsonville, South Carolina
  - Spartanburg, South Carolina
  - Dallas, Texas
  - Friendswood, Texas
  - Houston, Texas
  - Irving, Texas
  - Katy, Texas
  - Missouri City, Texas
  - North Richland Hills, Texas
  - Pearland, Texas
  - Sugarland, Texas
  - Riverton, Utah
  - Salt Lake City, Utah
  - Arlington, Virginia
  - Burke, Virginia
  - Manassas, Virginia
  - Port Orchard, Washington
- Puerto Rico (4):
  - Aguas Buenas
  - Aibonito
  - Loíza
  - San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 74 investigative sites in Puerto Rico and the United States from 30 October 2007 to 30 April 2009.
Pre-assignment Details: Black participants with essential hypertension were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Azilsartan Medoxomil 40 mg QD: Azilsartan medoxomil 40 mg, tablets, orally, once daily for up to 6 weeks.
- Azilsartan Medoxomil 80 mg QD: Azilsartan medoxomil 80 mg, tablets, orally, once daily for up to 6 weeks.
- Placebo QD: Azilsartan medoxomil placebo-matching tablets, orally, once daily for up to 6 weeks.
Period: Overall Study
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Started | 140 (Randomized or Treated) | 137 (Randomized or Treated) | 138 (Randomized or Treated)
Completed | 126 | 116 | 123
Not Completed | 14 | 21 | 15
Not completed — Adverse Event | 3 | 3 | 1
Not completed — Protocol Violation | 2 | 2 | 2
Not completed — Lost to Follow-up | 2 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 7 | 6
Not completed — Lack of Efficacy | 1 | 0 | 3
Not completed — Other | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD | Total
Number analyzed (Participants) | 138 | 137 | 138 | 413
Age Categorical [Number; unit: participants]
  <45 years | 29 | 37 | 36 | 102
  Between 45 and 64 years | 94 | 86 | 85 | 265
  ≥65 years | 15 | 14 | 17 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 80 | 78 | 236
  Male | 60 | 57 | 60 | 177

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the 24-hour Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -7.70 (1.063) | -10.48 (1.026) | -2.70 (1.065)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented. Overall 0.05 level of significance for multiple comparisons controlled using closed testing procedure; Mean Difference (Final Values) = -5.00, 95% CI 2-sided [-7.97 to -2.04]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.78, 95% CI 2-sided [-10.69 to -4.86]

2. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Systolic Blood Pressure
Description: The change in mean trough clinic sitting systolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 134 | 130 | 133
mmHg | -9.51 (1.330) | -9.58 (1.351) | -3.04 (1.333)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.48, 95% CI 2-sided [-10.18 to -2.78]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.54, 95% CI 2-sided [-10.27 to -2.81]

3. Secondary Outcome: Change From Baseline in the 24-hour Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in 24-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 24-hour mean is the average of all measurements recorded for 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -4.93 (0.732) | -7.27 (0.706) | -1.49 (0.731)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.001, ANCOVA — Postbaseline P-value was from ANCOVA with terms for treatment (as a factor) and baseline value (as a covariate). Unadjusted p-value is presented; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-5.47 to -1.40]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.77, 95% CI 2-sided [-7.78 to -3.77]

4. Secondary Outcome: Change From Baseline in Mean Trough Clinic Sitting Diastolic Blood Pressure
Description: The change in mean trough clinic sitting diastolic blood pressure measured at final visit or week 6 relative to baseline.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 134 | 130 | 133
mmHg | -5.48 (0.755) | -5.32 (0.766) | -2.36 (0.757)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.12, 95% CI 2-sided [-5.22 to -1.02]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -2.96, 95% CI 2-sided [-5.08 to -0.84]

5. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -7.53 (1.094) | -10.40 (1.056) | -2.43 (1.096)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.09, 95% CI 2-sided [-8.14 to -2.04]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.97, 95% CI 2-sided [-10.96 to -4.97]

6. Secondary Outcome: Change From Baseline in Daytime (6am to 10 pm) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in daytime (6am to 10pm) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Daytime mean is the average of all measurements recorded between the hours of 6 am and 10 pm.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -5.08 (0.764) | -7.24 (0.738) | -1.34 (0.764)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-5.86 to -1.61]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.90, 95% CI 2-sided [-7.99 to -3.81]

7. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -7.97 (1.303) | -10.34 (1.259) | -3.06 (1.307)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.91, 95% CI 2-sided [-8.54 to -1.27]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.27, 95% CI 2-sided [-10.85 to -3.69]

8. Secondary Outcome: Change From Baseline in the Nighttime (12 am to 6 am) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in nighttime (12am to 6am) mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. Nighttime mean is the average of all measurements recorded between the hours of 12 am and 6 am.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -4.48 (0.950) | -7.23 (0.916) | -1.44 (0.950)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.024, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.05, 95% CI 2-sided [-5.69 to -0.40]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.79, 95% CI 2-sided [-8.39 to -3.19]

9. Secondary Outcome: Change From Baseline in the 12-hr Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -7.70 (1.155) | -10.11 (1.114) | -2.40 (1.156)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.30, 95% CI 2-sided [-8.52 to -2.08]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.71, 95% CI 2-sided [-10.88 to -4.55]

10. Secondary Outcome: Change From Baseline in the 12-hr Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in the 12-hour mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The 12-hour mean is the average of all measurements recorded in the first 12 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -5.15 (0.815) | -6.99 (0.788) | -1.34 (0.816)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -3.81, 95% CI 2-sided [-6.08 to -1.54]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -5.65, 95% CI 2-sided [-7.88 to -3.41]

11. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Systolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean systolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -7.14 (1.382) | -10.99 (1.334) | -2.28 (1.385)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.014, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.86, 95% CI 2-sided [-8.72 to -1.01]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -8.71, 95% CI 2-sided [-12.50 to -4.92]

12. Secondary Outcome: Change From Baseline in the Trough (22-24-hr) Mean Diastolic Blood Pressure Measured by Ambulatory Blood Pressure Monitoring.
Description: The change in trough mean diastolic blood pressure measured at week 6 relative to baseline. Ambulatory blood pressure monitoring measures blood pressure at regular intervals throughout the day and night. The trough mean is the average of all measurements recorded from 22 to 24 hours after dosing.
Time Frame: Baseline and Week 6.
Population: Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 94 | 101 | 94
mmHg | -4.77 (1.126) | -8.28 (1.085) | -0.73 (1.125)
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.012, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -4.04, 95% CI 2-sided [-7.17 to -0.91]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -7.55, 95% CI 2-sided [-10.63 to -4.48]

13. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Systolic Blood Pressure Response, Defined as < 140 mm Hg and/or Reduction From Baseline ≥ 20 mm Hg
Description: Percentage of participants who achieve a clinic systolic blood pressure response measured at week 6, defined as less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Systolic blood pressure is the arithmetic mean of the 3 trough sitting systolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 134 | 130 | 133
percentage of participants | 41.8 | 37.7 | 24.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.004, Regression, Logistic — P-value for response criteria for systolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 2.15, 95% CI 2-sided [1.27 to 3.65]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.016, Regression, Logistic — [p-value comment as in outcome 13, analysis 1]; Odds Ratio (OR) = 1.93, 95% CI 2-sided [1.13 to 3.31]

14. Secondary Outcome: Percentage of Participants Who Achieve a Clinic Diastolic Blood Pressure Response, Defined as < 90 mm Hg and/or Reduction From Baseline ≥ 10 mm Hg
Description: Percentage of participants who achieve a clinic diastolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg. Diastolic blood pressure is the arithmetic mean of the 3 trough sitting diastolic blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 134 | 130 | 133
percentage of participants | 53.0 | 55.4 | 39.8
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.018, Regression, Logistic — P-value for response criteria for diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic diastolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 1.85, 95% CI 2-sided [1.11 to 3.08]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.015, Regression, Logistic — [p-value comment as in outcome 14, analysis 1]; Odds Ratio (OR) = 1.89, 95% CI 2-sided [1.13 to 3.16]

15. Secondary Outcome: Percentage of Participants Who Achieve Both a Clinic Diastolic and Systolic Blood Pressure Response
Description: Percentage of participants who achieve both a clinic diastolic and systolic blood pressure response measured at week 6, defined as less than 90 mm Hg and/or reduction from baseline of greater than or equal to 10 mm Hg AND less than 140 mm Hg and/or reduction from baseline of greater than or equal to 20 mm Hg. Diastolic and systolic blood pressure is based on the arithmetic mean of the 3 sitting blood pressure measurements.
Time Frame: Baseline and Week 6.
Population: Full analysis set with last observation carried forward.
Measure: Number; unit: percentage of participants
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Number analyzed (Participants) | 134 | 130 | 133
percentage of participants | 32.1 | 34.6 | 16.5
Statistical Analysis 1: Comparison: Azilsartan Medoxomil 40 mg QD vs Placebo QD; Test type: Superiority or Other; p = 0.004, Regression, Logistic — P-value for joint response criteria for systolic blood pressure and diastolic blood pressure was from a logistic regression with treatment as a factor and baseline clinic systolic blood pressure as a covariate. The unadjusted p-value is presented; Odds Ratio (OR) = 2.35, 95% CI 2-sided [1.31 to 4.24]
Statistical Analysis 2: Comparison: Azilsartan Medoxomil 80 mg QD vs Placebo QD; Test type: Superiority or Other; p < 0.001, Regression, Logistic — [p-value comment as in outcome 15, analysis 1]; Odds Ratio (OR) = 2.84, 95% CI 2-sided [1.57 to 5.13]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious adverse event) after the last dose of double-blind study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Azilsartan Medoxomil 40 mg QD | Azilsartan Medoxomil 80 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 3/137 | 1/137 | 0/138
Other Adverse Events (participants affected / at risk) | 6/137 | 9/137 | 3/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=137) | Azilsartan Medoxomil 80 mg QD (N=137) | Placebo QD (N=138)
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Azilsartan Medoxomil 40 mg QD (N=137) | Azilsartan Medoxomil 80 mg QD (N=137) | Placebo QD (N=138)
Headache (Nervous system disorders) | 6 | 9 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.